CLINICAL TRIAL: NCT01925248
Title: Can Whey Protein Improve Glycemic Control in Type 2 Diabetes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 474534; A-13-001-UCD-SK-NH (Other Grant/Funding Number: California Dairy research Foundation)
Record Dates: First submitted 2013-07-31; First posted 2013-08-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus; Hyperglycemia
Keywords: Whey protein; protein supplement; Diabetes; Type 2 DM; Hyperglycemia; Insulin secretagogue
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey protein group (Active Comparator): Patients will be randomized to receive whey protein
  Interventions: Dietary Supplement: Whey protein
- Placebo group (Placebo Comparator): Patients will be randomized to receive placebo
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Whey protein — Whey protein group participants will take supplement drinks that contain whey protein, daily before breakfast and before dinner for 3 months.
  Arms: Whey protein group
Dietary Supplement: Placebo group — Placebo group participants will take supplement drinks that do not contain whey protein, daily before breakfast and before dinner for 3 months.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate whether intake of protein supplement just before meals lowers the blood sugar levels after the meals. It is believe that pre-meal administration of a high-protein supplement can effectively improve glycemic control in type 2 diabetes (DM).

DETAILED DESCRIPTION:
11.3% of the population aged 20 years or older (25.6 million individuals) has diabetes. In the population aged 65 years or older, the prevalence of diabetes reaches to 26.9%.

Type 2 DM is caused by insulin resistance accompanied by insufficient compensatory insulin response. Therefore insulin secretagogues are a significant component of the therapeutic armamentarium. Insulin secretagogues, such as sulphonylureas and meglitinides, are routinely prescribed to lower post prandial glucose levels in type 2 DM. However, these medications are cleared by the liver and the kidneys and cannot be used in the presence of relevant co-morbidities. These medicines can also cause side effects, including hypoglycemia. Limitations of these medicines are likely to lead diabetic patients and their health care providers to seek alternate methods to treat postprandial hyperglycemia. Thus, our research which aims to identify an alternate insulin secretagogue is important and timely.

Whey protein (WP), a rich source of essential and branch chain (BC) amino acids (AA), is a potent insulin secretagogue. Although it is well known that protein and/or AA intakes stimulate insulin secretion, protein supplements are not being used clinically in order to lower post-prandial glycemia. WP can be a satisfactory alternative to the pharmaceutical insulin secretagogues.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 DM; age: 25 to 70y; BMI: 25 - 40 kg/m2; on no drug treatment or on metformin alone; HgBA1 6.5 - 8.5%; urinary microalbumin < 30 mg/g cr.

Exclusion Criteria:

* Systemic disease (liver, renal, untreated hypothyroidism, etc); in the last 2 mo: > 5% weight change, smoking, alcohol intake > 4 /wk; restricted diets; medications or herbals affecting insulin secretion/sensitivity . Pregnant women, prisoners, individuals who cannot provide informed consent.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Level | each day up to 3 months

SECONDARY OUTCOMES:
Change in 24 hour urine C-peptide excretion level | baseline and 1 month up to 3 months
Change in Weight | 1 month up to 3 months
Change in Body Mass Index (BMI) | 1 month up to 3 months
Change in vital signs | 1 month up to 3 months
Change in DEXA | baseline and 1 month up to 3 months
Change in Free fatty acids (FFA) levels | baseline and 1 month up to 3 months
Change in Lipid levels | baseline and 1 month up to 3 months
Change in GLP-1 levels | baseline and 1 month up to 3 months
Change in hs-CRP levels | baseline and 1 month up to 3 months
Change in Glycated hemoglobin (HgBA1C) level | baseline and 1 month up to 3 months
Change in Urine glucose level | baseline and 1 month up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sidika E Kasim-Karakas, M.D., Principal Investigator — University of California, Davis
Locations (1):
- Clinical and Translational Science Center Clinical Resources Center (CCRC), Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No